CLINICAL TRIAL: NCT05980832
Title: The Effect of Peer Education-Supported Psychosocial Skills Education Applied to Individuals With Chronic Mental Disorder on Patients' Perceptions of Stigma, Levels of Functionality and Insight
Brief Title: Effect of Peer-Supported Psychosocial Skills Training in Individuals With Chronic Mental Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halil İbrahim Bilkay, Psychiatric Nurse, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TOGU-HEM-HİB-01
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Mental Disorders; Peer Support; Psychosocial Skills Training; Functionality; Stigmatization; Insight
MeSH Terms: conditions — Stereotyping

STUDY DESIGN:
Masking Description: Masking could not be done in the study because training was to be provided. The identification and randomization of groups will be performed by the center staff using the blinding technique without the knowledge of the researcher to avoid bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group 1 (Experimental): It will consist of 10 patients who have received psychosocial skills training by the staff of the center, and a 6-week peer-supported psychosocial skills training will be given by the peer-leaders trained by the researcher psychiatric nurse.
  Interventions: Other: Peer Education Supported Psychosocial Skills Education
- Experimental Group 2 (Experimental): It will consist of 10 patients who have not received psychosocial skills training by the staff of the center, and a 6-week peer-supported psychosocial skills training will be given by the peer-leaders trained by the researcher psychiatric nurse.
  Interventions: Other: Peer Education Supported Psychosocial Skills Education
- Control Group 1 (No Intervention): It will consist of 10 patients who have received psychosocial skills training by the center staff and no intervention will be applied.
- Control Group 2 (No Intervention): It will consist of 10 patients who have not received psychosocial skills training by the center staff and no intervention will be applied.
- Peer Practitioner Training (Other): It is the group in which psychosocial skills training will be given to 4 patients with chronic mental disorders by a researcher psychiatric nurse.
  Interventions: Other: Peer practitioner training - Peer Education Supported Psychosocial Skills Education

INTERVENTIONS:
Other: Peer practitioner training - Peer Education Supported Psychosocial Skills Education — Psychosocial skills training-practitioner training will be given to 4 patients diagnosed with chronic mental disorder by the research psychiatry nurse.
  Educational content
  1. Getting acquainted - briefing about the study
  2. The Importance, Aims and Objectives of Psychosocial Skills Education
  3. The importance of peer support
  4. The importance, aims and objectives of peer education supported psychosocial skills training
  5. Management of the meeting game, warm-up games and role plays
  6. 1st and 2nd session peer education supported psychosocial skills training
  7. 3rd and 4th session peer education supported psychosocial skills training
  8. The last 5th and 6th sessions of peer education are supported by psychosocial skills training.
  9. Key points and termination in group management. The training will be planned to last 10-13 hours in total. Trainer's booklet prepared by the researcher psychiatric nurse.
  Arms: Peer Practitioner Training
Other: Peer Education Supported Psychosocial Skills Education — It is a psychosocial skills training that will be given to both experimental groups in 6 sessions within 6 weeks. 2 of the 4 peer trainers who received the practitioner training will conduct the training. During the training period, the research psychiatric nurse will support.
  Session titles are as follows:
  1. Session:Preparation Session
  2. Session: Understanding Mental Disorders
  3. Session: Developing Communication Skills
  4. Session: Developing Emotion Recognition and Expression Skills
  5. Session: Dealing with Daily Living Activities and Problems
  6. Session: Understanding the Stigma Experience
  The duration of each session is determined as 90 minutes. Taking into account the patient's opinions breaks not exceeding 15 minutes will be given as needed.
  Arms: Experimental Group 1; Experimental Group 2

SUMMARY:
This study was designed to examine the effects of peer education-supported psychosocial skills training on stigma perceptions, social functionality and insight levels of chronic psychiatric patients followed up in a community mental health center.

The research was planned as a mixed method study conducted in a randomized controlled experimental study design and a qualitative study design. With the findings obtained, it is aimed to increase the social functionality of the patients, to increase the level of insight and to reduce the perception of stigma, and to close an important gap in the literature, thanks to peer education-supported psychosocial skills training.

DETAILED DESCRIPTION:
Hypothesis(s) and Question(s):

The hypotheses of the quantitative method of the research are as follows; H1-1: Peer Education Supported Psychosocial Skills Training has an effect on the social functionality levels of patients.

H1-2: Peer Education Supported Psychosocial Skills Training has an effect on patients' perceptions of stigma.

H1-3: Peer Education Supported Psychosocial Skills Training has an effect on patients' insight levels.

The research questions of the qualitative method of the research are as follows:

Q(1): How do the changes experienced by people with chronic mental disorders affect their lives? Q(2): How does Peer Education Supported Psychosocial Skills Training affect patients' social functionality levels? Q(3): How does Peer Education Supported Psychosocial Skills Training affect patients' perceptions of stigma? Q(4): How does Peer Education Supported Psychosocial Skills Training affect patients' insight levels? Q(5): What are the experiences and opinions of the patients who participated in the Peer Education Supported Psychosocial Skills Training program?

The research question created for the research to be mixed method:

Q(Mixed): Do the themes revealed by the statements of the patients as a result of the qualitative research support the quantitative findings obtained as a result of the quantitative research?

Data Collection and Intervention

Firstly, A 13-hour practitioner training about psychosocial skills training supported by peer education and group management will be given by the research psychiatric nurse to 4 patients (one as peer leader, other as assistant, the other two as substitutes) selected according to the inclusion criteria of the study.

Individuals who are called peer trainers and who are subjected to practitioner training by the researcher psychiatric nurse will carry out the 6-session psychosocial skills training as leaders and assistant leaders. Researcher psychiatric nurse will support them in this process, even if they need it. It is thought that with the education given by peer educators, patients can benefit from each other's experiences and have an effect on the relevant variables. Groups will be determined by lot by the center staff from among the patients who have or have not received psychosocial skills training before.

In the research, "Descriptive Information Form" will be used by the researcher as a data collection tool, indicating the sociodemographic characteristics of the participants. The measurement of the variables specified in the research will be provided by the Self Stigma Scale, Beck Cognitive Insight Scale and Social Functioning Assessment Scale.

In order to evaluate the qualitative data, a semi-structured interview form consisting of questions about the effectiveness of education on the variables will be used by the researcher. After the pre-test application, a measurement will be made at the end of the sessions in the 2nd week, 4th week and 6th week in order to measure the effectiveness of the study during the application. Also, a measurement will be made in the 8th week for follow-up purposes.

After the collection of quantitative data, 5 people from both experimental groups will be selected and qualitative data will be collected with 10 participants in total. Individual and face-to-face interviews will be conducted with the patients who make up the experimental group, and the interviews will be audio recorded with the knowledge and consent of the participant. Individual interviews will be provided with a semi-structured form for the effectiveness of the training.

ELIGIBILITY:
Inclusion Criteria:

For peer practitioner training:

* Being registered with the Community Mental Health Center (CMHC),
* Participating in the study voluntarily and being an instructor in 6 sessions of psychosocial skills training.
* Having a high level of functionality according to the functionality scale
* Not in the active period of the disease
* Being able to read and write and not have any communication problems in understanding and speaking Turkish.
* Well-being for at least 6 months according to the treatment team and according to the records.

For Peer-Supported Psychosocial Skills Training:

* Coming to CMHC regularly
* Volunteer to participate in the study and agree to attend 6-week sessions
* Not in the active period of the disease.
* Ability to read, write and communicate in Turkish
* Being healthy for at least 6 months according to the treatment team and records
* Having the experience of receiving standard psychosocial skills training by mental health professionals working in the institution for Experimental Group 1 and Control Group 1.
* Not having received standard psychosocial skills training by the mental health professionals working in the institution for Experiment Group 2 and Control Group 2 are the inclusion criteria determined for peer educator-supported psychosocial skills training.

Exclusion Criteria:

* Not registering with CMHC.
* Inability to give written informed consent to the study
* Inability to communicate in written or verbal Turkish at a level that will complete the assessments and be included in the groups.
* The emergence of acute illness symptoms during the education process
* The conflict between the patient giving the training and the patients participating in the group training constitutes the exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Functionality (Social Functioning Assessment Scale) | 6 Weeks
  This scale evaluates 19 items and four sub-dimensions in general in patients with schizophrenia. Among the factors, interpersonal explanations and entertainment consist of seven items, self-care seven items, independent living needs four items, and work-life one item. The scores that can be obtained from the scale are between 19 and 57, and a high score means that social functioning measures are high.
  It is expected that there will be an increase in the functionality levels of the experimental groups.
Stigmatization (Self-Stigma Scale) | 6 Weeks
  It is a 3-factor scale consisting of 17 items for patients evaluating self-stigmatization or internalized stigma, concealment of illness and perception of worthlessness in individuals with mental illness. A five-point Likert-type scale was created as "1=not at all suitable for me, 2=somewhat appropriate, 3=moderately appropriate, 4=generally appropriate, 5=completely appropriate". As the score obtained from the scale increases, the self-stigmatization of the patients increases. The Cronbach's alpha correlation coefficient value of the scale is 0.93, indicating high reliability.
  It is expected that the stigma perceptions of the experimental groups will decrease.
Insight (Beck Cognitive Insight Scale) | 6 Weeks
  The Turkish validity and reliability study of the scale developed to assess cognitive insight was conducted. The scale, which is a four-point Likert type, consists of 15 items and has 2 sub-dimensions "self-confidence" and "self-evaluation". The scoring system of the scale consists of "disagree" 0 points, "somewhat agree" 1 point, "mostly agree" 2 points, "strongly agree" 3 points. The total (composite) score of the scale is obtained by subtracting the self-evaluation items (1,3,4,5,6,8,12,14,15) from the self-confidence item scores (2,7,9,10,11,13). The total score range of the scale is between -18 and 27 points. A high score indicates a high level of insight. In the reliability study of the Turkish version of the scale, the internal consistency Cronbach's alpha coefficient was found to be 0.68.
  It is expected that there will be an increase in the insight levels of the experimental groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Gürhan, Prof. Dr., Study Director — Tokat Gaziosmanpa University
Locations (1):
- Samsun Mental Health and Diseases Hospital - Community Mental Health Center, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The identity information of the participants will not be shared with other researchers. The statistical data of the research is planned to be published in a scientific journal.